CLINICAL TRIAL: NCT02382146
Title: A Prospective Randomize Study: Prevention of Nausea and Vomiting in Plastic Surgery
Brief Title: Prevention of Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, nurcan kizilcik, Dr., Yeditepe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: yeditepe universty hospital
Record Dates: First submitted 2015-02-24; First posted 2015-03-06 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexamethasone and ondansetron (Experimental): dexamethasone 8 mg with ondansetron 4mg administered in group DO
  Interventions: Drug: dexamethasone ondansetron
- dexamethasone and dimenhydrinate (Active Comparator): dexamethasone 8 mg with dimenhydrinate 1mg/kg administered in group DD
  Interventions: Drug: Dexamethasone dimenhidrinate

INTERVENTIONS:
Drug: dexamethasone ondansetron — dexamethasone 8 mg intravenous ondansetron 4 mg intravenous dimenhydrinate 1mg/kg intravenous
  Other Names: dekort zofer dramamine
  Arms: dexamethasone and ondansetron
Drug: Dexamethasone dimenhidrinate — dexamethasone 8 mg intravenous dimenhydrinate 1mg/kg intravenous
  Other Names: dekort dramamin
  Arms: dexamethasone and dimenhydrinate

SUMMARY:
We designed this randomized, double- blind, single-center study to compare the efficacy of the combination of dexamethasone with ondansetron and dexamethasone with dimenhydrinate undergoing plastic surgery.

DETAILED DESCRIPTION:
A total of 60 voman patient, ASA status I-II , aged 18-65 year and scheduled for elective rhinoplasty were enrolled in the study. Exclusion criterias hypersensitivity or contraindication for the studied medications, received an antiemetic drug or steroid within 24 hours before anesthesia, have history of diabetes history of motion sickness (MS) or PONV, or pregnant and lactating females.

Patients were informed on how to use the patient controlled analgesia device during the postoperative period. The risk criterias for PONV were recorded for each patient.Patients were randomly assigned to two study groups of 30 patients. All patients were premedicated with intravenous (iv) midazolam (1-2 mg). On arrival in the operating room, standard anesthetic monitors were applied. Anesthesia was induced with iv propofol (2-3 mg/kg) and fentanyl (1-1.5 μg/kg). Tracheal intubation was facilitated with rocuronium (0.6 mg/kg). After tracheal intubation all patient received iv 8 mg dexamethasone. Normocapnic mechanical ventilation was performed after intubation. General anesthesia was maintained with sevoflurane (1 minimum alveolar concentration) in oxygen / air mixture and remifentanil (0.1-0.3 μg/kg/min) infusion.Four mg ondansetron and for each patient 1 mg/kg dimenhydrinate in the 5 ml syringe solution were prepared by pharmacy department, and given to the blinded investigators. The patients, anesthesiologists (with the exception of the primary author), statistician, and observes were all blinded.

Dimenhydrinate was administered in group DD (1mg/kg), and ondansetron was administered in group DO (4mg), and all patients received tramadol (1.5mg/kg) and tenoksikam (20mg) half an hour before emergence.

Postoperative analgesia was provided with a patient controlled analgesia system by using iv tramadol (5mg/mL) (2 ml bolus and 10 minutes lockout interval without basal infusion).

After the surgery, muscle relaxation was reversed by administering neostigmine (0.05mg/kg) and atropine (0.015mg/kg). Patients were extubated and transferred to the recovery unit.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

18 Years to 60 Years woman

ASA (American Society of Anesthesiologist) physical status I or II

Patients undergoing laparoscopic gynecologic surgery or laparoscopic cholecystectomy

Exclusion Criteria:

Hypersensitivity or contraindication to the study medications,

Antiemetic drug or steroid use within 24 hours before anesthesia,

History of diabetes mellitus,

History of motion sickness or postoperative nausea and vomiting,

Pregnancy,

Breast feeding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
prevention of postoperative nausea and vomiting | 1 year
  The primary outcome is complete response: complete response is defined as no postoperative nausea (VRS≤3), retching or vomiting and no need for rescue antiemetic.

CONTACTS AND LOCATIONS:
Overall Officials: nurcan kızılcık, Principal Investigator — yeditepe UH
Locations (1):
- Turkey, Istanbul, Kadıkoy, Turkey (Türkiye)